CLINICAL TRIAL: NCT06045546
Title: A (5-5-5-8) Technique for Laparoscopic Cholecystectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ClinAmygate (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR00C1947
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cholecystitis; Gallstone; Cholecystolithiasis; Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Gallstones; Cholecystolithiasis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-5-5-8 group (Experimental): In this group, the new 5-5-5-8 technique of laparoscopic cholecystectomy will be done.
  Interventions: Procedure: 5-5-5-8 technique
- Control (Active Comparator): In this group, the 10-10-5-5 technique of laparoscopic cholecystectomy will be done.
  Interventions: Procedure: 10-10-5-5 technique

INTERVENTIONS:
Procedure: 5-5-5-8 technique — the new technique of 5-5-5-8 for laparoscopic cholecystectomy
  Arms: 5-5-5-8 group
Procedure: 10-10-5-5 technique — the standard technique of 10-10-5-5 for laparoscopic cholecystectomy
  Arms: Control

SUMMARY:
The aim of this current study is to investigate the effectiveness and safety of a novel technique which is the 5-5-5-8 where the camera port is 5 mm.

DETAILED DESCRIPTION:
More than 50 different LC procedures are described in the literature, mostly as a result of changes made by surgeons to enhance cosmetic and postoperative results. Some adjustments include port size and/or number reductions relative to conventional LC usage. Each of these methods has benefits and drawbacks, and each one is appropriate for usage in particular circumstances.

The aim of this current study is to investigate the effectiveness and safety of a novel technique which is the 5-5-5-8 where the camera port is 5 mm.

The study has two analyses:

1. at 6 month follow up
2. at 24 months follow up

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patients eligible for LC during the study period

Exclusion Criteria:

* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Duration of the operation | 1 hour
  Duration of the operation in minutes
Number of participants with Conversion to open surgery | 1 hour
  Number of participants with Failure of the technique and conversion to open surgery
Incidence of intra operative visceral injury | 2 hours
  Incidence of intra operative visceral injury
intra operative amount of blood loss | 2 hours
  intra operative amount of blood loss in ml
incidence of intra operative complications | 2 hours
  incidence of intra operative complications

SECONDARY OUTCOMES:
post operative stay | 1 week
  post operative stay in days
incidence of port site infection | 1 month
  incidence of infection of the port site
Incidence of port site hernia | 6 months
  Incidence of hernia of the port site
Incidence of port site hernia | 12 months
  Incidence of hernia of the port site
Incidence of port site hernia | 24 months
  Incidence of hernia of the port site

CONTACTS AND LOCATIONS:
Overall Officials: Mohie El-Din M Madani, MD, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be shared after approval of the IRB